CLINICAL TRIAL: NCT03723499
Title: Feasibility and Therapeutic Method of Endoscopic Treatment of Bronchial Carcinoid Tumors: 22 Years Experience of Saint-Etienne
Brief Title: Endoscopic Treatment of Bronchial Carcinoid Tumors
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN812018/CHUSTE
Record Dates: First submitted 2018-10-26; First posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Carcinoid Tumor
Keywords: Carcinoid tumors; Endoscopic treatment; Recurrence
MeSH Terms: conditions — Carcinoid Tumor; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- endoscopic treatment: Patient with endoscopic treatment will be included. Some medical data collection by medical record will be collected.
  Interventions: Other: Medical data collection

INTERVENTIONS:
Other: Medical data collection — Medical data collection by medical record will be collected: demographics data, medical history, clinical symptoms, smoking, type of endoscopic method, complete treatment or not, type of surgeries if yes, anatomopathology of the injury and recurrence if yes

SUMMARY:
Carcinoid tumors of the lung are considered to be a low-grade malignancy. Surgical resection is considered the standard approach. Recent data has shown that a complete endoscopic treatment could be considered. An endoscopic treatment is can be a alternative to invasive surgery.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the feasibility and therapeutic method of endoscopic treatment of bronchial carcinoid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated by endoscopic approach for a carcinoid tumor at the University Hospital Centre of Saint-Etienne between November 1995 to December 2017.

Exclusion Criteria:

* Patients treated for a recurrence of carcinoid tumor.
* Patients with metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by endoscopic approach for a carcinoid tumor will be included.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 1995-11 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Complete endoscopic treatment | Month 1
  patients who have a complete endoscopic treatment

SECONDARY OUTCOMES:
Type of endoscopic method used | Month 1
  Analysis type of endoscopic method used.
Tumor localization | Month 1
  Analysis the tumor localization.
Deadline before recurrence | 10 years
  Analysis the deadline before recurrence of the tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel VERGNON, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No